CLINICAL TRIAL: NCT06764862
Title: A Randomised, Double-blind, Placebo-controlled Parallel Group Phase II Clinical Study Evaluating the Efficacy and Safety of HSK44459 Tablets in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Evaluating the Efficacy and Safety of of HSK44459 in People With Idiopathic Pulmonary Fibrosis
Acronym: IPF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK44459-201
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK44459-dose 1 (Experimental)
  Interventions: Drug: HSK44459 dose 1
- HSK44459-dose 2 (Experimental)
  Interventions: Drug: HSK44459 dose 2
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK44459 dose 1 — HSK44459 taken orally twice daily in the morning and in the evening for 12 weeks.
  Arms: HSK44459-dose 1
Drug: HSK44459 dose 2 — HSK44459 taken orally twice daily in the morning and in the evening for 12 weeks.
  Arms: HSK44459-dose 2
Drug: Placebo — Placebo matching HSK44459 taken orally twice daily in the morning and in the evening for 12 weeks.
  Arms: Placebo

SUMMARY:
This study is open to adults with idiopathic pulmonary fibrosis who are at least 40 years old. The main objective is to evaluate of the efficacy and the secondary objective is to evaluate the safety and pharmacokinetic.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Idiopathic Pulmonary Fibrosis (IPF) prior to screening, patients must meet both of the following criteria:

1. IPF based on 2022 ATS/ERS/JRS/ALAT Guideline as confirmed by the investigator based on chest HRCT scan taken before or during screening period and if available surgical lung biopsy.
2. Usual interstitial pneumonia (UIP) or probable UIP HRCT pattern consistent with the clinical diagnosis of IPF, as confirmed by the investigator prior to screening. if indeterminate HRCT finding IPF may be confirmed locally by (historical) biopsy.

2. Percentage Predicted Forced Vital Capacity (ppFVC) ≥45% at screening period. 3. Diffusion capacity of the lung for carbon monoxide (DLCO) (corrected for haemoglobin [Hb]) ≥ 25% of predicted normal at screening period.

4. Patients have to be either:

1. not on therapy with nintedanib or pirfenidone for at least 8 weeks prior to screening and during the screening period, and not planning to start or restart anti fibrotic therapy.
2. on stable therapy with nintedanib or pirfenidone for at least 8 weeks prior to screening and during the screening period.

Exclusion Criteria:

1. Clinically significant airways obstruction (Forced Expiratory Volume in One Second (FEV1)/Forced Vital Capacity (FVC) < 0.7) at screening.
2. In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
3. Acute IPF exacerbation within 4 months prior to screening and/or during the screening period (investigator-determined).
4. Lower respiratory tract infection requiring antibiotics within 2 weeks prior to screening and/or during the screening period.
5. Major surgery (major according to the investigator's assessment) performed within 3 months prior to screening or planned during the course of the trial. (Being on a transplant list is allowed).
6. History of malignancy within 5 years prior to screening.
7. Any suicidal behavior within 2 years prior to screening (i.e. actual attempts, interrupted attempts, abandoned attempts, or prepared actions or attitudes).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-27 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in forced vital capacity (FVC) at week 12 | day 1 and week 12
  FVC is a standard pulmonary function test used to quantify respiratory muscle weakness

SECONDARY OUTCOMES:
Relative change from baseline in FVC at week 12 | day 1 and week 12
  FVC is a standard pulmonary function test used to quantify respiratory muscle weakness
The change from baseline in percentage predicted forced vital capacity ( ppFVC) at week 12 | day 1 and week 12
  FVC is a standard pulmonary function test used to quantify respiratory muscle weakness